CLINICAL TRIAL: NCT01494948
Title: Innate Immunity and the Allergic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 221035-2
Record Dates: First submitted 2011-11-07; First posted 2011-12-19 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Nasal Allergies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): skin test negative
  Interventions: Other: allergen challenge
- allergic (Active Comparator): Skin test positive
  Interventions: Other: allergen challenge

INTERVENTIONS:
Other: allergen challenge — nasal challenges with antigen to which they are sensitive to

SUMMARY:
The purpose of this study is to determine if a certain cell type (the CD49d+ neutrophil) is associated with the presence or development of allergic disease.

DETAILED DESCRIPTION:
A specific subset of neutrophils (CD49d+) will be recruited to the nasal tissue of individuals with allergic disease, and that these cells will also be found in the peripheral blood of allergic subjects. Normal subjects (those without atopy) and those treated for atopic disease will lack the presence of these cells.

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent before any study related activity is performed
2. Male and female adult and adolescent patients aged ≥18 years and ≤ 65 years.
3. Allergic or non-allergic subjects as proven by allergy skin tests in the past 2 years.

Exclusion Criteria:

1. The presence of any of these diseases: Atopic dermatitis, persistent controlled asthma, any level of severity of uncontrolled asthma, immunodeficiency or suspected immunodeficiency, any co-morbid disease (cardiac, congenital, diabetes, renal, gastrointestinal, hematologic, and oncologic).
2. Any prior history of immunodeficiency, cardiac, congenital, diabetes, renal, gastrointestinal, hematologic, or oncologic disease.
3. The use of any intranasal and inhaled corticosteroids within the last month.
4. Current therapy with any medication other than as needed over-the-counter medications or as-needed (not scheduled) antihistamine use.
5. Current pregnancy.
6. Women of childbearing potential not using an acceptable birth control method, as well as women who are breastfeeding
7. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (specify as required)
8. Use of any other investigational agent in the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Increase in percentage of CD49d expressing neutrophils in nasal lavage post allergen challenge. | 1month
  Nasal lavage on atopic and non-atopic adult subjects will be performed at baseline and following an allergen challenge. The frequency of CD49d expressing neutrophils in the lavage fluid will be determined by flow cytometry analysis, and the change in this frequency will be correlated with atopic status and allergen challenge. This is an observational study, procedures performed are not intended to impact the outcome of the individual participants.

SECONDARY OUTCOMES:
Change in immune cell numbers in the nasal lavage following allergen challenge | 1 month
  The numbers of neutrophils, CD49d+ neutrophils, lymphocytes, dendritic cells, and macrophages in the nasal lavage will be determined before and after allergen challenge. The outcome will be correlation of these changes with allergy status and any clinical symptoms of the allergen challenge (i.e., sneezing).

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Grayson, MD, Principal Investigator — Medical College of Wisconsin

REFERENCES:
- [Result] Sigua JA, Buelow B, Cheung DS, Buell E, Hunter D, Klancnik M, Grayson MH. CD49d-expressing neutrophils differentiate atopic from nonatopic individuals. J Allergy Clin Immunol. 2014 Mar;133(3):901-4.e5. doi: 10.1016/j.jaci.2013.09.035. Epub 2013 Dec 18. No abstract available. PMID 24360325